CLINICAL TRIAL: NCT01722240
Title: Liraglutide in Type 1 Diabetes
Acronym: 1966
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Paresh Dandona, Director, Diabetes-Endocrinology Center of Western NY, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1966; 1R01DK092653-01A1 (NIH)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide 1.8mg (Active Comparator): Daily Injection
  Interventions: Drug: Liraglutide 1.8mg
- Placebo (Placebo Comparator): Daily Injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide 1.8mg
  Arms: Liraglutide 1.8mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The glucose lowering effects of GLP-1 agonists are well established in subjects with type 2 diabetes, however, these have not been studied prospectively in subjects with type 1 diabetes. The investigators have, therefore, designed this study to investigate the central hypothesis that in patients with type 1 diabetes, Liraglutide has a glucose lowering effect. A major secondary objective of this study is to elucidate the mechanisms responsible for its glucose lowering effects and those involved in reducing the insulin dose. The specific aims of this proposal are:

Hypothesis 1: Treatment with Liraglutide in patients with type 1 diabetes decreases HbA1c, fasting, postprandial and the overall mean glucose concentrations while decreasing the dose of insulin required.

Hypothesis 2: Treatment with Liraglutide in patients with type 1 diabetes decreases basal and postprandial glucagon concentrations and increases basal and postprandial C-peptide concentrations.

Hypothesis 3: Treatment with Liraglutide in patients with type 1 diabetes delays gastric emptying.

DETAILED DESCRIPTION:
The control of glucose homeostasis in subjects with type 1 diabetes is fragile since exogenous insulin cannot compensate for changing requirements and is not precise either in terms of the dose or the bio-availability of the insulin injected. Furthermore, in the near total absence of insulin secretion, the physiological post prandial inhibition of glucagon secretion by the α-cell is also probably deficient in all type 1 diabetics. Thus, there is a need for therapies beyond insulin that can further improve glycemic control and reduce fluctuations in glucose in these subjects. The investigators have recently shown that Liraglutide, a glucagon like peptide (GLP)-1 analogue with duration of action of 24 hours, when added to insulin in subjects with well controlled type 1 diabetes reduces mean and standard deviation of blood glucose, HbA1c and insulin requirements. Since C-peptide concentrations did not alter following Liraglutide, it is likely that the suppression of glucagon may have contributed to this effect. The glucose lowering effects of GLP-1 agonists are well established in subjects with type 2 diabetes, however, these have not been studied prospectively in subjects with type 1 diabetes. The investigators have, therefore, designed this study to investigate the central hypothesis that in patients with type 1 diabetes, Liraglutide has a glucose lowering effect. A major secondary objective of this study is to elucidate the mechanisms responsible for its glucose lowering effects and those involved in reducing the insulin dose. The specific aims of this proposal are:

Hypothesis 1: Treatment with Liraglutide in patients with type 1 diabetes decreases HbA1c, fasting, postprandial and the overall mean glucose concentrations while decreasing the dose of insulin required.

Aim 1.1: To compare the HbA1c, mean fasting, glucose, mean weekly glucose, standard deviation of weekly blood glucose concentrations as recorded by continuous glucose monitoring and the dose of insulin required prior to and following 52 weeks of treatment with 1.8 mg of liraglutide daily.

Aim 1.2: To compare the postprandial glucose concentrations following a test meal before and after 52 weeks of treatment with 1.8 mg of liraglutide daily.

Hypothesis 2: Treatment with Liraglutide in patients with type 1 diabetes decreases basal and postprandial glucagon concentrations and increases basal and postprandial C-peptide concentrations.

Aim 2.1: To compare the basal and postprandial glucagon and C-peptide concentrations following a test meal before and after 52 weeks of treatment with 1.8 mg of liraglutide daily.

Hypothesis 3: Treatment with Liraglutide in patients with type 1 diabetes delays gastric emptying.

Aim 3.1: To compare the gastric emptying as measured by acetaminophen absorption before and after treatment with 1.8 mg of daily subcutaneous liraglutide.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 Diabetes on continuous subcutaneous insulin infusion (CSII; also known as insulin pump) or multiple (four or more) injections of insulin per day.
2. Regularly measuring blood sugars four times daily.
3. HbA1c of less than 8.5%.
4. Well versed with carbohydrate counting.
5. Age 18-75 years.
6. BMI 20-40 kg/m2

Exclusion Criteria:

1. Type 1 diabetes for less than 6 months;
2. Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks;
3. Hepatic disease (transaminase > 3 times normal) or cirrhosis;
4. Renal impairment (serum eGFR < 30ml/min/1.73m2);
5. HIV or Hepatitis B or C positive status;
6. Participation in any other concurrent clinical trial;
7. Any other life-threatening, non-cardiac disease;
8. Use of an investigational agent or therapeutic regimen within 30 days of study.
9. history of pancreatitis
10. pregnancy
11. inability to give informed consent
12. history of gastroparesis
13. history of medullary thyroid carcinoma or MEN 2 syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MBBS, PhD, Principal Investigator — Kaleida Health
Locations (1):
- Diabetes-Endocrinology Center of WNY, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Exclusion Criteria: Type 1 diabetes for less than 6 months. Coronary event or procedure (myocardial infraction, unstable angina, coronary artery bypass surgery or coronary angioplasty) in the previous four weeks. Hepatic disease (transamine > 3 times normal) or cirrhosis. Renal impairment (serum eGFR < 30 mL/min/1.73m2).
Groups:
- Liraglutide: Liraglutide 1.8 mg Daily Injection
- Placebo: Daily placebo Injection
  Placebo
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 35 | 34
Completed | 26 | 20
Not Completed | 9 | 14

BASELINE CHARACTERISTICS:
Population: Out of 69 patients enrolled in the study, 13 patients dropped out from the study before baseline/randomization visit (during the 30 days insulin dose optimization).
  Therefore, baseline data is from 29 and 27 patients only.
Groups:
- Liraglutide 1.8mg: Daily Injection
  Liraglutide 1.8mg
- Placebo: Daily Injection
  Placebo
- Total: Total of all reporting groups
Arm/Group | Liraglutide 1.8mg | Placebo | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 45 (2) | 47 (3) | 46 (2.5)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: male and female counted here as a separate category
  Participants
    Gender: male | 12 | 14 | 26
    Gender: female | 17 | 13 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
HbA1c (%) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 7.92 (0.19) | 7.50 (0.18) | 7.71 (0.18)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 28.9 (1.1) | 29.1 (1.6) | 29.0 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c (%)
Description: HbA1c measured at baseline and after 52 weeks of treatment with Liraglutide or placebo.
Time Frame: 52 Weeks
Measure: Mean (Standard Error); unit: Percent of Hemoglobin (%)
Groups:
- Liraglutide: Daily Injection
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 26 | 20
Percent of Hemoglobin (%)
  week 0 | 7.92 (0.15) | 7.48 (0.18)
  week 52 | 7.45 (0.12) | 7.58 (0.14)

2. Secondary Outcome: Mean Weekly Glucose Concentrations.
Description: Mean weekly glucose concentrations measured by CGM at baseline and at 52 weeks
Time Frame: 52 Weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 26 | 20
mg/dL
  week 0 | 173 (5) | 160 (6)
  week 52 | 156 (6) | 156 (6)

3. Secondary Outcome: Body Weight
Description: Body weight in Kg measured at weeks 0 (baseline) and at 52 weeks after treatment with liraglutide or placebo
Time Frame: 52 weeks
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 26 | 20
Kg
  week 0 | 83.6 (3.8) | 84.1 (4.0)
  week 52 | 80.5 (3.8) | 83.8 (4.0)

ADVERSE EVENTS:
Time Frame: 56 weeks
Description: Safety data is collected for 56 weeks (4 weeks before randomization and 52 after randomization)
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/20
Other Adverse Events (participants affected / at risk) | 0/26 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT01722240/Prot_SAP_000.pdf